CLINICAL TRIAL: NCT03209024
Title: App Documentation of Electronic BP Readings in Hypertension
Brief Title: Smartphone App Assisted Home Blood Pressure Monitoring Amongst Hypertensive Patients in Singapore
Acronym: ADELPHY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: SingHealth Polyclinics (Other)
Responsible Party: Principal Investigator, Professor Tazeen Jafar, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017/2014
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Hypertension
Keywords: hypertension; home blood pressure monitoring; self blood pressure monitoring; telemedicine; health apps; informatics; data collection; personal health records; smartphone; self care; blood pressure monitors
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: open, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Participants complete a 3-week home blood pressure monitoring regimen using a handwritten logbook to record all blood pressure readings.
  Interventions: Other: Handwritten logbook recording of home blood pressure readings
- Intervention (Experimental): Participants complete a 3-week home blood pressure monitoring regimen using a smartphone app and Bluetooth® technology to wirelessly record all blood pressure readings.
  Interventions: Device: Smartphone assisted wireless recording of home blood pressure readings

INTERVENTIONS:
Other: Handwritten logbook recording of home blood pressure readings — Participants use a handwritten logbook to record the details of their home blood pressure measurements, including systolic blood pressure, diastolic blood pressure, date, and time.
  Arms: Control
Device: Smartphone assisted wireless recording of home blood pressure readings — Participants use a smartphone app and Bluetooth® technology to wirelessly record the details of their home blood pressure measurements, including systolic blood pressure, diastolic blood pressure, date, and time.
  Arms: Intervention

SUMMARY:
Background: Hypertension is the leading attributable risk factor for cardiovascular disease and death globally. In diagnosing and monitoring hypertensive patient population, home blood pressure monitoring (HBPM) has been shown to be superior to the office-based blood pressure (BP) measurement as a predictor of cardiovascular disease and total mortality. However, the conventional method of HBPM utilizing handwritten BP logbooks has known shortcomings, mainly attributable to inaccuracy and underreporting of data, as well as the failure to bring the logbooks to the regular outpatient appointments. In recent years, the availability of home BP devices with Bluetooth® technology on the market, the increasingly widespread use of smartphones, and the development of mobile applications (apps) that complement Bluetooth® enabled BP monitors have expanded the potential for an accurate log of BP data to be accessible to clinicians. Our study's primary aim is to compare the level of HBPM recording fidelity using smartphone app versus using a handwritten logbook among the multi-ethnic hypertensive patient population seen in a district polyclinic located in Pasir Ris, Singapore. Patient acceptability of the two recording modalities and the association between the home blood pressure recording fidelity and the patients' socio-demographic background, self-care profile, clinical factors, and level of exposure to technology is also assessed as exploratory aims. Our main hypothesis is that the level of fidelity in HBPM recording, defined as the proportion of scheduled number of home blood pressure readings that is successfully recorded, regimen compliant, and made available at the final follow up visit, would be higher for patients who use a smartphone app versus those who maintain a handwritten logbook.

Methods/design: Open, randomized controlled trial of 80 patients seen at Pasir Ris Polyclinic randomized to either intervention or control arm and assessed after a 3-week follow up period

Intervention arm: Participants randomized to intervention arm follow a 3-week HBPM regimen and wirelessly record the BP readings onto a smartphone app using Bluetooth® technology.

Control arm: Participants randomized to control arm follow a 3-week HBPM regimen (identical to intervention arm) and manually record the BP readings onto a handwritten logbook.

Participants: A convenience sample of 80 patients visiting the study polyclinic was obtained during the recruitment period (15 Mar 2017 - 15 June 2017).

Outcomes: A trained outcomes assessor will assess each participant's home BP record brought to the final follow up visit at 3 weeks post-randomization. The primary outcome will be HBPM recording fidelity, defined as the proportion of scheduled number of home blood pressure readings that is successfully recorded, regimen compliant, and made available at the final follow up visit. The participants' level of discomfort during the study, their willingness to incorporate into their healthcare management the modality of HBPM to which they were assigned, and their overall impression on their study participation will be assessed by a participant acceptability questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Singaporean citizen or permanent resident
* Able to communicate in English
* Diagnosis of essential hypertension and on at least one antihypertensive medical therapy
* Between 40-70 years of age
* Owns a smartphone compatible with the study
* Has been visiting the study polyclinic for at least 1 year

Exclusion Criteria:

* Known cardiac arrhythmia
* Known end stage renal disease
* Known cancer patient
* Known history of stroke
* Known history of myocardial infarct
* Physical or mental disability that would prevent one's own measurement of home BP (e.g. visual impairment, dementia)
* Maximal arm circumference exceeding BP cuff size
* Anticipation of extensive travel overseas during study period
* Occupation requires night shift
* Participating in other clinical trials

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-07-31 (Estimated); Study Completion 2017-07-31 (Estimated)

PRIMARY OUTCOMES:
Home Blood Pressure Recording Fidelity within each study arm | Baseline visit to 3 weeks post randomization
  The proportion of scheduled number of home blood pressure readings that is successfully recorded, regimen compliant, and made available at the final follow up visit.

SECONDARY OUTCOMES:
The association of participants' age with home blood pressure recording fidelity within each study arm | Baseline visit to 3 weeks post randomization
  regression coefficient p-value < 0.05 is considered to be statistically significant
The association of participants' highest level of education with home blood pressure recording fidelity within each study arm | Baseline visit to 3 weeks post randomization
  regression coefficient p-value < 0.05 is considered to be statistically significant
The association of participants' years of smartphone use with home blood pressure recording fidelity within each study arm | Baseline visit to 3 weeks post randomization
  regression coefficient p-value < 0.05 is considered to be statistically significant

OTHER OUTCOMES:
Participant Acceptability of the home blood pressure recording modality within each study arm | Baseline visit to 3 weeks post randomization
  A trained outcomes assessor administers the Participant Acceptability Questionnaire to assess the participants' level of discomfort during the study, their willingness to incorporate into their healthcare management the modality of HBPM to which they were assigned, and their overall impression on their study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen Jafar, MD, MPH, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- SingHealth Polyclinics - Pasir Ris, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawes CM, Vander Hoorn S, Rodgers A; International Society of Hypertension. Global burden of blood-pressure-related disease, 2001. Lancet. 2008 May 3;371(9623):1513-8. doi: 10.1016/S0140-6736(08)60655-8. PMID 18456100
- [Background] Niiranen TJ, Hanninen MR, Johansson J, Reunanen A, Jula AM. Home-measured blood pressure is a stronger predictor of cardiovascular risk than office blood pressure: the Finn-Home study. Hypertension. 2010 Jun;55(6):1346-51. doi: 10.1161/HYPERTENSIONAHA.109.149336. Epub 2010 Apr 12. PMID 20385970
- [Background] Mengden T, Hernandez Medina RM, Beltran B, Alvarez E, Kraft K, Vetter H. Reliability of reporting self-measured blood pressure values by hypertensive patients. Am J Hypertens. 1998 Dec;11(12):1413-7. doi: 10.1016/s0895-7061(98)00241-6. PMID 9880121
- [Background] Stergiou GS, Baibas NM, Gantzarou AP, Skeva II, Kalkana CB, Roussias LG, Mountokalakis TD. Reproducibility of home, ambulatory, and clinic blood pressure: implications for the design of trials for the assessment of antihypertensive drug efficacy. Am J Hypertens. 2002 Feb;15(2 Pt 1):101-4. doi: 10.1016/s0895-7061(01)02324-x. PMID 11863243
- [Background] Ohkubo T, Asayama K, Kikuya M, Metoki H, Hoshi H, Hashimoto J, Totsune K, Satoh H, Imai Y; Ohasama Study. How many times should blood pressure be measured at home for better prediction of stroke risk? Ten-year follow-up results from the Ohasama study. J Hypertens. 2004 Jun;22(6):1099-104. doi: 10.1097/00004872-200406000-00009. PMID 15167443
- [Background] Chatellier G, Day M, Bobrie G, Menard J. Feasibility study of N-of-1 trials with blood pressure self-monitoring in hypertension. Hypertension. 1995 Feb;25(2):294-301. doi: 10.1161/01.hyp.25.2.294. PMID 7843782
- [Background] Tamaki S, Nakamura Y, Teramura M, Sakai H, Takayama T, Okabayashi T, Kawashima T, Horie M. The factors contributing to whether or not hypertensive patients bring their home blood pressure record to the outpatient clinic. Intern Med. 2008;47(18):1561-5. doi: 10.2169/internalmedicine.47.0710. Epub 2008 Sep 16. PMID 18797113
- [Background] Han HR, Lee H, Commodore-Mensah Y, Kim M. Development and validation of the Hypertension Self-care Profile: a practical tool to measure hypertension self-care. J Cardiovasc Nurs. 2014 May-Jun;29(3):E11-20. doi: 10.1097/JCN.0b013e3182a3fd46. PMID 24088621
- [Background] Wu H, Wang B, Zhu X, Chu G, Zhang Z. A new automatic blood pressure kit auscultates for accurate reading with a smartphone: A diagnostic accuracy study. Medicine (Baltimore). 2016 Aug;95(32):e4538. doi: 10.1097/MD.0000000000004538. PMID 27512876
- [Background] Tinetti ME, Han L, Lee DS, McAvay GJ, Peduzzi P, Gross CP, Zhou B, Lin H. Antihypertensive medications and serious fall injuries in a nationally representative sample of older adults. JAMA Intern Med. 2014 Apr;174(4):588-95. doi: 10.1001/jamainternmed.2013.14764. PMID 24567036
- [Derived] Moon EW, Tan NC, Allen JC, Jafar TH. The Use of Wireless, Smartphone App-Assisted Home Blood Pressure Monitoring Among Hypertensive Patients in Singapore: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 May 28;7(5):e13153. doi: 10.2196/13153. PMID 30905872